CLINICAL TRIAL: NCT01589679
Title: Contracture Reduction Following Bunionectomy: a Longitudinal, Controlled Trial
Acronym: Bunionectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unrelated to Trial
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DYN1-12-047
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Hallux Limitus
MeSH Terms: conditions — Hallux Limitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control/ standard of care (Other): ALL SUBJECTS WILL RECEIVE SHOE INSERTS AND HOME STRETCHING REGIME. Control subjects will be treated with the Standard of Care during the first 12 weeks, but after the 12 weeks patients will be fit with MTP, which delivers a low-load, prolonged-duration stretch after completion of this study.
  Interventions: Other: standard of care
- Dynasplint (Experimental): ALL SUBJECTS WILL RECEIVE SHOE INSERTS AND HOME STRETCHING REGIME. Experimental subjects will be immediated treated with the Metatarsal Dynasplint, which delivers a low-load, prolonged-duration stretch for 60 minutes, three times per day.
  Interventions: Device: Metarsal Dynasplint

INTERVENTIONS:
Other: standard of care — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. This unit is work for 60 minutes three times per day.
  Arms: control/ standard of care
Device: Metarsal Dynasplint — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. This unit is work for 60 minutes three times per day.
  Arms: Dynasplint

SUMMARY:
To determine the efficacy of Metatarsal Dynasplint Sytem (MTP) in reducing contracture of hallux limitus secondary to Bunionectomy, in a longitudinal, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis 1st MTJ Contracture following Bunionectomy

Exclusion Criteria:

* Current treatment with Botulinium Toxin-A (Botox), lower extremity
* Current treatment Fluoroquinolones (antibiotic medication)
* Current use of muscle relaxant medications
* Fibromyalgia
* Stroke, CVA, Brain Injury, Spinal Cord Injury, or any neural pathology causing plasticity or hypertonicity
* Treatment with electrical stimulation assisting ambulation (i.e Bioness, WalkAide, Parastep, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
A Repeated Measures Analysis of Variance (ANOVA) | 12 months
  ANOVA will be performed to measure different in category, pain, duration to full restoration of active range of motion(AROM).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - Brown Hand Center and Achilles Foot & Ankle Specialist, Henderson, Nevada
  - Advanced Diagnostic Foot and Ankle Specialist of Cy-Fair, Houston, Texas